CLINICAL TRIAL: NCT01237639
Title: Transfusion of Red Cells in Hematopoietic Stem Cell Transplantation: The TRIST Study
Brief Title: Study of Red Blood Cell Transfusion Triggers in Patients Undergoing Hematopoietic Stem Cell Transplantation
Acronym: TRIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Blood Services (Other); Canadian Institutes of Health Research (CIHR) (Other Government); The Ottawa Hospital (Other); Hamilton Health Sciences Corporation (Other); London Health Sciences Centre (Other); Saskatchewan Cancer Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20120673
Record Dates: First submitted 2010-10-13; First posted 2010-11-09 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hematologic Malignancies
Keywords: Red Cells; Transfusion; Trigger; Threshold; Hematopoietic Stem cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive Red blood cell Transfusion (Experimental): Transfusion Trigger of 70g/L with an aim to maintain Hemoglobin between 80-90g/L
  Interventions: Other: Red blood cell Transfusion
- Liberal Red blood Cell Transfusion (Active Comparator): Transfusion Trigger of 90g/L with an aim to maintain Hemoglobin between 100-110g/L
  Interventions: Other: Red blood cell Transfusion

INTERVENTIONS:
Other: Red blood cell Transfusion — Transfusion of Red blood cells to based on daily complete blood count

SUMMARY:
Transfusion of red blood cells (RBCs) is important for the care of patients undergoing stem cell transplantation. Stem cell transplants are used to treat blood cancers and bone marrow disorders. This involves the use of high doses of chemotherapy and/or radiation to kill cancer cells; but this damages the marrow and blood system. Blood stem cells are transplanted by infusing into the recipient and blood counts recover over 2-3 weeks. Before bone marrow recovery, RBCs are needed to support the patient. Higher hemoglobin in these high risk patients may have benefits such as better energy and organ function. However, research in other areas of medicine suggests that a higher red cell count may be dangerous. Taken together, it is unclear whether having a lower or higher red cell count is better for patients having a blood stem cell transplant. The investigators plan to study this by randomly assigning patients having a transplant to be transfused with RBCs either at a higher or lower hemoglobin level. In this way, the investigators will be able to accurately find out if there are any benefits or harms in having a lower or higher red cell count during the recovery period after blood stem cell transplantation.

DETAILED DESCRIPTION:
1. Males or females aged 18 years or older who are undergoing either an autologous or allogeneic HSCT.
2. The indications for HSCT may include, but not limited to the following diseases :

   1. Acute Leukemia, myeloid, lymphoid or biphenotypic in 1st, 2nd remission or in relapse
   2. Chronic Myeloid Leukemia in chronic, accelerated or blast phase
   3. Chronic Lymphocytic Leukemia
   4. Myelodysplastic Syndrome
   5. Myeloproliferative Disorder
   6. Lymphoma
   7. Myeloma
3. All study patients must provide consent at least 1 day prior to scheduled HSCT and provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 16-70 undergoing either an autologous or allogeneic HSCT for any hematologic malignancy

Exclusion Criteria:

* Pregnant or lactating at the time of enrollment
* Already received red cell transfusion after HSCT but prior to enrollment
* Unable/unwilling to provide informed consent.
* Patients receiving HSCT for non-malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QOL)/Function based on the FACT-BMT scale | 3 years
  The FACT consists of 5 subscales that measure physical well-being, functional well-being, social/family well-being and emotional well-being. The BMT subscale of the FACT includes additional items specifically designed to test quality of life and symptoms specific to BMT patients.

SECONDARY OUTCOMES:
Transplant Related Mortality | 100 days
Red Cell Transfusion | 100 days
Platelet Transfusion | 100 days
Acute Graft Versus Host Disease | 100 days
Bleeding | 100 days
  Grade 3 or 4 by WHO scale
Serious Infections | 100 days
  All grade 4 and 5 infections (according to the CTCAE v.4)
Time to Non-relapse Mortality | 100 days
Economic Evaluation/Quality of Life | 100 days
  EQ-5D
NCI Toxicity Scale | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tay, MD FRCPC MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Saskatchewan Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Tay J, Tinmouth A, Fergusson D, Allan D. Transfusion of red cells in hematopoietic stem cell transplantation (TRIST): study protocol for a randomized controlled trial. Trials. 2011 Sep 21;12:207. doi: 10.1186/1745-6215-12-207. PMID 21936907
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Tay J, Allan DS, Chatelain E, Coyle D, Elemary M, Fulford A, Petrcich W, Ramsay T, Walker I, Xenocostas A, Tinmouth A, Fergusson D. Liberal Versus Restrictive Red Blood Cell Transfusion Thresholds in Hematopoietic Cell Transplantation: A Randomized, Open Label, Phase III, Noninferiority Trial. J Clin Oncol. 2020 May 1;38(13):1463-1473. doi: 10.1200/JCO.19.01836. Epub 2020 Feb 21. PMID 32083994